CLINICAL TRIAL: NCT00728676
Title: Pilot Study to Evaluate the Effects of Kuvan on Adult Individuals With Phenylketonuria With Measurable Maladaptive Behaviors
Brief Title: Study to Evaluate the Effects of Kuvan on Individuals With Phenylketonuria (PKU) With Maladaptive Behaviors
Status: Completed | Type: Observational
Sponsor: Shoji Yano (Other)
Collaborators: BioMarin Pharmaceutical (Industry)
Responsible Party: Sponsor-Investigator, Shoji Yano, Director, Genetics Division,, University of Southern California
Organization: University of Southern California (Other)
Other Study IDs: BioMarin-300
Record Dates: First submitted 2008-07-30; First posted 2008-08-06 (Estimated); Last update posted 2013-01-18 (Estimated); Status verified 2013-01

CONDITIONS: Phenylketonuria
Keywords: PKU,; Phe,; PAH,; Kuvan,; Trp,; Tyr
MeSH Terms: conditions — Phenylketonurias

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
To validate the outcome measures and the tolerability of Kuvan treatment in the improvement of behavioral symptoms in 10 selected adults with Phenylketonuria (PKU) with or without mental retardation.

ELIGIBILITY:
Inclusion Criteria:

* Biochemical confirmation of PKU,
* Measurable maladaptive behavior at baseline,
* Signed informed consent,
* Not pregnant or lactating,
* Females on birth control if applicable,
* Willing to comply.

Exclusion Criteria:

* Subjects or care provider unreliable, use of investigational products within 30 days prior to enrollment,
* Pregnant or lactating,
* Concurrent disease or condition that would interfere with study participation or safety, ie multiple psychotropic meds, any condition the PI renders the subject at high risk, on drugs that inhibit folate synthesis,
* Concurrent use of levodopa.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Individuals with PKU followed at our clinic
Sampling Method: Non-Probability Sample
Enrollment: 10 (Actual)
Dates: Start 2008-08; Primary Completion 2010-03 (Actual); Study Completion 2010-05 (Actual)

PRIMARY OUTCOMES:
Pattern of change from baseline to 6 and 12 months in Vineland scale standard scores, evaluated with a repeated measure ANOVA approach. | One year

SECONDARY OUTCOMES:
Correlation and regression methods (non-linear if appropriate) to examine the relationship between changes in behavior and in amino acid profiles. | one year

CONTACTS AND LOCATIONS:
Overall Officials: Shoji Yano, MD, Ph.D., Principal Investigator — University of Southern California
Locations (1):
- LAC+USC Medical Center, Los Angeles, California, United States